CLINICAL TRIAL: NCT02402374
Title: Randomized, Placebo-controlled, Blind-assessor Study to Evaluate the Safety and Efficacy of Autologous Platelet Rich Plasma Gel Prepared With the RegenKit-BCT Plus Family of Kits for the Treatment of Diabetic Foot Ulcer
Brief Title: Evaluate the Safety and Efficacy of RegenKit Autologous PRP Gel for the Treatment of Diabetic Foot Ulcer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Regen Lab SA (Industry)
Collaborators: RegenLab USA LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014-WH-02
Record Dates: First submitted 2015-03-25; First posted 2015-03-30 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2019-12

CONDITIONS: Diabetic Foot Ulcers
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- PRP gel (Experimental): Autologous platelet rich plasma gel
  Interventions: Device: Autologous platelet rich plasma gel
- Placebo (Placebo Comparator): Saline gel
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Autologous platelet rich plasma gel — PRP gel application to exuding wounds, such as leg ulcers, pressure ulcers, and diabetic foot ulcers and for the management of mechanically- or surgically-debrided wounds
  Arms: PRP gel
Device: Placebo — Placebo control arm will be receiving commercial formulations of pre-prepared saline gel.
  Arms: Placebo

SUMMARY:
Autologous platelet-rich plasma (PRP) gel was reported to have very good outcomes in the treatment of foot ulcers in pilot studies and retrospective uncontrolled trials. Therefore, a larger randomized, placebo-controlled clinical trial will be useful to determine whether platelet-rich plasma is safe and effective for the treatment of diabetic foot ulcers (DFU).

DETAILED DESCRIPTION:
Evaluate the safety and efficacy of RegenKit autologous PRP Gel for the treatment of diabetic foot ulcer is a randomized, placebo controlled, blind-assessor study. One hundred and seventy four patients will be treated, 87 patients receiving treatment arm and 87 patients receiving placebo. The primary endpoint is to evaluate proportion of patients with complete wound closure at week 16 when treated with autologous platelet rich plasma gel compared to the proportion of control (saline gel) treated patients with complete wound closure at the same time-point.

ELIGIBILITY:
Inclusion Criteria

* Patients who in the opinion of the Investigator, are capable of understanding and complying with protocol requirements
* Patients or, when applicable, their legal representatives, sign and dates a written IFC and/or any required privacy authorization prior to the initiation of any study procedure
* Patients aged 18 to 95 (inclusive) with Type 1 or Type 2 diabetes undergoing therapy for glycemic control
* Patients with glycated hemoglobin (HbA1C) less than or equal to 12%
* Patients having ulcers which meet the following criteria:
* Ulcer should not be infected as determined by clinical examination
* Ulcer duration of 4 weeks or longer
* Ulcer area (length x width) of between 1.5 cm2 and 20 cm2
* Full-thickness ulcer of Grade 1 or Grade 2 as per Wagner's classification system
* Ulcer has undergone recent debridement (2 weeks prior to screening)
* Post-debridement ulcer is free of necrotic debris, foreign bodies, sinus tracts, tunneling, and undermining and is comprised of healthy vascularized tissue
* Patients with Charcot deformity, the wound should be free of acute changes and, in the opinion of Investigator, should have undergone appropriate structural consolidation (the affected charcot fractures will have been fused together and should be sufficiently stable to allow the patient to weight-bear)
* Patients having adequate circulation to the foot as documented by either:

  1. Ankle Brachial Index (ABI) between 0.60 and 1.30, or
  2. Patients with falsely elevated ABI values (equal to or greater than 1.30) due to non-compressible ankle vessels:

  i)Toe Brachial Index (TBI) equal to or greater than 0.50 or, ii)TBI is not available (toe is absent, wounds are present, or investigative site cannot perform a TBI), a Doppler waveform in the posterior tibial or dorsalis pedis arteries at the ankle consistent with adequate flow in the foot (biphasic or triphasic) and other diagnostic confirmation of adequate flow (e.g duplex imaging or normal pulse volume recording)
* Patients who agree to conform to the off-loading requirements
* Patients of childbearing age must agree to use a method of contraception or agree to abstain from sexual intercourse throughout the study

Exclusion Criteria

* Patients with ulcers having an active infection with/without purulent discharge
* Patients with ulcers with exposed bone or associated with osteomyelitis
* Patients with target limb cellulitis, or ischemic or gangrenous ulcers
* Patients who have undergone, in the 2-week period prior to enrollment, treatment for DFU with any advanced treatment modality other than standard of care, such as growth factors, skin substitutes or other biological treatments
* Female patients who are pregnant or lactating
* Patients diagnosed with cancer, undergoing chemotherapy, except basal cell carcinoma
* Patients with wounds caused by basal cell carcinoma or due to basal cell carcinoma excision
* Patients with wounds due to malignancy
* Patients having had any revascularization surgery within the 4-week period prior to signing the ICF
* Patients with renal failure requiring dialysis
* Patients with platelet count outside of the normal range of 150-400 x 1000/uL
* Patients with a history of allergy to one of tested components
* Patients with a history of bleeding disorders
* Patients suffering from skin or blood cancers, or having suffered in the past from such cancers and not having, certification of a total remission
* Patients presenting skin lesions potentially caused by abnormal cellular proliferation process (history of being cancerous)
* Patients with a history of any condition, physical examination finding, or clinical laboratory finding, giving reasonable suspicion of a disease or condition that contraindicates the use of the investigational agent or may confound the interpretation of study results or might render the patient at high risk for treatment complications
* Patients with active Charcot or other structural deformity that would prevent adequate off-loading of the study foot

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2018-04-12 (Actual); Primary Completion 2020-10-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with complete wound closure | 16 weeks
  Proportion of patients with complete wound closure at week 16 when treated with autologous platelet rich plasma gel compared to the proportion of control (saline gel)-treated patients with complete wound closure at the same time-point.

CONTACTS AND LOCATIONS:
Overall Officials: Alisha Oropallo, MD, Principal Investigator — Northwell Health, Comprehensive Wound Care Center
Locations (1):
- Futuro Clinical Trials, McAllen, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
The Institution and the Principal Investigator are free to publish, present, or use any data and results arising out of this Study, provided that such publication does not disclose any of Sponsor's Confidential Information. Sponsor shall be able to present data and results at symposia, national or regional professional meetings, and publish in journals, theses or dissertations, or otherwise of its own choosing. In the event that the Principal Investigator fails to submit a formal academic publication within twelve (12) months following completion of the Study, the Sponsor is entitled to prepare a publication based on the data and results. Such proposed publication will be submitted to the Institution for review and comment at the least thirty (30) calendar days before submission for publication.